CLINICAL TRIAL: NCT04861532
Title: Development of Protocols and Methods for Image Processing and Enhancement of MRI Data
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Collaborators: Medic Vision Imaging Solutions (Unknown)
Responsible Party: Sponsor
Other Study IDs: 0106-16-HYMC
Record Dates: First submitted 2021-04-14; First posted 2021-04-27 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-04

CONDITIONS: MRI Image Enhancement
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: Imaging — MRI scanning using new protocols

SUMMARY:
The purpose of the study is to develop new Magnetic Resonance Imaging (MRI) protocols and methods for image processing and enhancement. Different setting of acquisition parameters used in conventional clinical MRI protocols will be defined, to create "New Protocols". Then post-processing will be applied on new protocols to enhance the image quality. Finally a comparison of image quality will be performed to compare the image quality of images obtained by conventional protocols with those obtained with the New Protocols.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers for clinical MRI examination
* Patients undergoing clinical MRI examination
* Capable to provide an informed written consent form

Exclusion Criteria:

* Any contraindication to MRI scanning, such as pacemakers or heart rhythm disturbances, permanent cosmetics or certain metallic implants in the body (excluding dental implants).
* Age <18 years old
* Pregnancy
* Claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Total number of subjects expected to participate in this study is up to 100. This study will be performed at multiple sites and data will be collected from different MRI scanners of variable field strength using several MRI protocols. To provide sufficient statistical power for the investigation of each subgroup, we need a large sample size.
  Children, pregnant women and prisoners that are considered vulnerable population by federal regulation will not be included in this study. In addition, decisional incapacity subject will be excluded.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Image Signal to Noise Ratio (SNR) | Through study completion, an average of 2 months.
  Comparing the SNR of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
Image Resolution | Through study completion, an average of 2 months.
  Comparing the resolution of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
Artifacts | Through study completion, an average of 2 months.
  Comparing artifacts of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
MRI contrast | Through study completion, an average of 2 months.
  Comparing MR contrast of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).
Diagnostic quality | Through study completion, an average of 2 months.
  Comparing diagnostic quality of images obtained by conventional protocols with the corresponding New Protocols' processed images. The comparison will be performed by neuroradiologists, using a 7-point Likert-scale. Where higher the score, better the outcome (1 means unacceptable and 7 means excellent).

CONTACTS AND LOCATIONS:
Overall Officials: Libi Mori, Study Director — Medic Vision Imaging Solutions Ltd; Roni Shreter, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe, Hadera, Select One, Israel

IPD SHARING:
Plan to Share IPD: Undecided